CLINICAL TRIAL: NCT00995436
Title: Efficiency and Effectiveness of Three Methods of Anchorage Reinforcement in Orthodontics
Brief Title: Chesterfield Micro-implant Study Involving Three Types of Anchorage Methods in Orthodontics
Acronym: PJSPhD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chesterfield and North Derbyshire Royal Hospital (Other Government)
Responsible Party: Principal Investigator, Jonathan Sandler, Principal Investigator, Chesterfield and North Derbyshire Royal Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07/Q2401/50; REC 07/Q2401/50 (Other: UK NHS Ethics); BOSF 2006 Grant 1 (Other Grant/Funding Number: British Orthodontics Foundation)
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Malocclusion; Class II Buccal Segment Relationship
Keywords: Extractions; Anchorage supplementation
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extraoral anchorage (Active Comparator): The intervention is the placement of Headgear, to be worn 100 hours per week
  Interventions: Device: Extraoral anchorage
- Miniscrews (Active Comparator): The intervention is the of miniscrews to supplement anchorage
  Interventions: Device: Miniscrews
- Nance palatal arch (Active Comparator): Anchorage supplemented by Nance palatal arch fixing molars together with an arch
  Interventions: Device: Nance

INTERVENTIONS:
Device: Extraoral anchorage — Extra oral anchorage
  Arms: Extraoral anchorage
Device: Miniscrews — Intraoral skeletal anchorage using mini screws
  Other Names: miniscrew for anchorage reinforcement
  Arms: Miniscrews
Device: Nance — Intraoral dental anchorage by using Nance palatal arch on molars
  Other Names: Nance button
  Arms: Nance palatal arch

SUMMARY:
Research problem:

Anchorage reinforcement is effective with headgear provided patient compliance is optimal. Nance palatal arch have also been shown to be effective. Microscrews despite their popularity however have no scientific evidence to support their use.

Aim:

To compare the effectiveness of 3 methods of anchorage reinforcement 1) headgear 2) Nance palatal arch 3) orthodontic micro-screws.

Hypothesis:

There is no difference in the amount of anchorage loss between the three methods of anchorage reinforcement.

Design:

Randomized clinical trial.

Setting: District General Hospital orthodontic department

Participants: 78 patients requiring "absolute anchorage".

Interventions: The subjects will be randomized into 3 groups. In group 1 headgear will be requested 12-14 hours per day. In group 2 a nance palatal arch will be placed for use as intra oral anchorage reinforcement. In group 3, orthodontic micro-screws will be used for anchorage.

Method of investigation:

The study will be of 78 'absolute anchorage' patients older than 12 years randomly assigned to one of three groups of anchorage reinforcement

Outcome measures:

1. Anchorage loss measured from lateral Cephalometric radiographs and 3-D model scanning, records will be taken at three points
2. Patient perception of the different treatment methods, including surgical experience

Data analysis: The data will be analysed on an intention to treat basis. Basic descriptive statistics and uni-variate tests will initially be done to explore the data. Final data analysis will involve the relevant multi-variate statistical modeling.

Dissemination: Conference proceedings, journal papers and the Cochrane oral health group.

DETAILED DESCRIPTION:
Research problem:

Anchorage reinforcement is effective with headgear provided patient compliance is optimal. Nance palatal arch have also been shown to be effective. Microscrews despite their popularity however have no scientific evidence to support their use.

Aim:

To compare the effectiveness of 3 methods of anchorage reinforcement 1) headgear 2) Nance palatal arch 3) orthodontic micro-screws.

Hypothesis:

There is no difference in the amount of anchorage loss between the three methods of anchorage reinforcement.

Design:

Randomized clinical trial.

Setting: District General Hospital orthodontic department

Participants: 78 patients requiring "absolute anchorage".

Interventions: The subjects will be randomized into 3 groups. In group 1 headgear will be requested 12-14 hours per day. In group 2 a nance palatal arch will be placed for use as intra oral anchorage reinforcement. In group 3, orthodontic micro-screws will be used for anchorage.

Method of investigation:

The study will be of 78 'absolute anchorage' patients older than 12 years randomly assigned to one of three groups of anchorage reinforcement

Data analysis: The data will be analysed on an intention to treat basis. Basic descriptive statistics and uni-variate tests will initially be done to explore the data. Final data analysis will involve the relevant multi-variate statistical modeling.

I took professional statistical advice from a senior statistician at the University of Manchester. Analysis of covariance was used and Headgear (as our default treatment) was used as the reference category. Results with Nance and TADs are relative to the reference category of headgear.

ELIGIBILITY:
Inclusion Criteria:

* Seventy-five children maximum anchorage cases, aged aged 12-17 referred from the General Dental Service to Chesterfield Royal Hospital will be selected to take part in this study.
* Informed consent will be obtained.

Exclusion Criteria:

* Previous orthodontic treatment,
* Unwillingness to accept any of the three methods of treatment, OR
* Syndromes or clefts.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2008-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sandler, BDSMSc MOrth, Study Chair — Chesterfield North Derbyshire NHS Trust
Locations (1):
- Chesterfield Royal Hospital, Chesterfield, Derbyshire, United Kingdom

REFERENCES:
- [Result] Sandler J, Murray A, Thiruvenkatachari B, Gutierrez R, Speight P, O'Brien K. Effectiveness of 3 methods of anchorage reinforcement for maximum anchorage in adolescents: A 3-arm multicenter randomized clinical trial. Am J Orthod Dentofacial Orthop. 2014 Jul;146(1):10-20. doi: 10.1016/j.ajodo.2014.03.020. PMID 24974994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted between August 2008 and February 2013 in two orthodontic departments in the United Kingdom.
Pre-assignment Details: 90 patients assesses as eligible. 12 chose not to take part
Groups:
- Headgear: Placement of extraoral traction to be worn 100 hours per week
  Extraoral anchorage : Extra oral anchorage using headgear
- Miniscrews: Placement of micro-screw to supplement anchorage
  Intraoral skeletal anchorage - Temporary anchorage device : Intraoral skeletal anchorage using mini screws
- Nance Palatal Arch: Anchorage supplemented by fixing molars together with an arch
  Intraoral dental anchorage : Intraoral dental anchorage by using Nance palatal arch on molars
Period: Overall Study
Arm/Group | Headgear | Miniscrews | Nance Palatal Arch
Started | 25 (25) | 27 | 26
Completed | 23 | 22 | 26
Not Completed | 2 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Headgear | Miniscrews | Nance Palatal Arch | Total
Number analyzed (Participants) | 25 | 27 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.38 (1.67) | 14.15 (1.25) | 14.14 (1.48) | 14.22 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 19 | 39
  Male | 15 | 17 | 7 | 39
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 27 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Anchorage Loss Measured From 3-D Model Scanning
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Miniscrews: Device Placement of micro-screw to supplement anchorage
  Intraoral skeletal anchorage - Temporary anchorage device: Intraoral skeletal anchorage using mini screws
- Nance Palatal Arch: Anchorage supplemented by fixing molars together with an arch
  Intraoral dental anchorage: Intraoral dental anchorage by using Nance palatal arch on molars
Arm/Group | Miniscrews | Nance Palatal Arch | Headgear
Number analyzed (Participants) | 22 | 26 | 23
mm
  Maxillary right molar | 0.80 (1.6) | 1.84 (1.32) | 1.36 (1.83)
  Maxillary left molar | 0.99 (1.15) | 2.09 (1.32) | 1.99 (2.09)
Statistical Analysis 1: Comparison: Miniscrews vs Headgear; Test type: Non-Inferiority or Equivalence — The calculation indicated that for a study with the power of 80% and an alpha of 0.05 we required 21 participants per group. Assumed drop out rate 20%, suggesting 75 patients required; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.53 to 0.36] — Maxillary right molar
Statistical Analysis 2: Comparison: Miniscrews vs Headgear; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.89 to -0.04] — Maxillary left molar
Statistical Analysis 3: Comparison: Nance Palatal Arch vs Headgear; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.32 to 1.55] — Maxillary right molar
Statistical Analysis 4: Comparison: Nance Palatal Arch vs Headgear; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1 to 0.83] — Maxillary left molar
Statistical Analysis 5: Comparison: Miniscrews vs Nance Palatal Arch vs Headgear; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, ANCOVA — Maxillary right molar. F(2, 67) = 3.10. Overall effect of treatment
Statistical Analysis 6: Comparison: Miniscrews vs Nance Palatal Arch vs Headgear; Maxillary left molar; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.08, ANCOVA — Overall effect of treatment F(2,67) = 2.58

2. Secondary Outcome: Patient Perception of the Different Treatment Methods, Including Surgical Experience
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Headgear: Device Placement of extraoral traction to be worn 100 hours per week
  Extraoral anchorage: Extra oral anchorage
Arm/Group | Headgear | Miniscrews | Nance Palatal Arch
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes